CLINICAL TRIAL: NCT05791838
Title: Borderline Ovarian Tumors: Results of a Retrospective, Single-center Experience
Brief Title: Experience in Borderline Ovarian Tumors
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Andrea Etrusco, Principal investigator, University of Palermo
Other Study IDs: BOT-1
Record Dates: First submitted 2023-02-08; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Borderline Ovarian Tumor
Keywords: Conservative surgery; Micropapillary patterns; Surgical staging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Borderline ovarian tumors (BOTs) comprise 15-20% of primary ovarian neoplasms and represent an independent disease entity among epithelial ovarian cancers. The present study aimed to report the 8-year experience of a single center on the management and outcomes of consecutive BOTs patients. From January 2010 to December 2017, all patients with BOTs undergoing surgical treatment were included. Demographic, clinical, and pathological data were reviewed retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years,
* Patients affected by borderline ovarian tumors (BOT) of any histological type and any FIGO stage,
* Women undergoing surgical treatment with both laparoscopic and laparotomic approaches.

Exclusion Criteria:

- Women affected by ovarian cancers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients surgically treated for borderline ovarian tumors (BOT)
Sampling Method: Non-Probability Sample
Enrollment: 86 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Oncological outcome | through study completion, an average of 1 year
  Patients who underwent surgery for BOT

CONTACTS AND LOCATIONS:
Overall Officials: Basilio Pecorino, M.D., Principal Investigator — University of Catania; Paolo Scollo, M.D. Ph.D., Study Director — University of Catania; Antonio Simone Laganà, M.D. Ph.D., Study Chair — University of Palermo; Andrea Etrusco, M.D., Study Chair — University of Palermo